CLINICAL TRIAL: NCT00226837
Title: Quantifying Nitrous Oxide Effect on Depth of Anaesthesia Using Theoretically Based Time Series Modelling
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: Australian and New Zealand College of Anaesthetists (Other)
Responsible Party: David Breeze, Cortical Dynamics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2004.109
Record Dates: First submitted 2005-09-26; First posted 2005-09-27 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Depth of Anaesthesia
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): 0% nitrous oxide
  Interventions: Drug: Nitrous oxide
- 2 (Active Comparator): 33% nitrous oxide
  Interventions: Drug: Nitrous oxide
- 3 (Active Comparator): 66% nitrous oxide
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Drug: Nitrous oxide — nitrous oxide by inhalation during induction
  Other Names: No other names were used

SUMMARY:
Our hypothesis is that a new method of depth of anaesthesia monitoring, using theoretically based time series modelling will result in improved ability to determine nitrous oxide anaesthetic effect

DETAILED DESCRIPTION:
We randomised patients to 0% 33% or 66% nitrous oxide during sevoflurane induction and measured anesthetic endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Presenting for surgery under general anaesthesia

Exclusion Criteria:

* Poor English language comprehension
* Risk of reflux
* Epilepsy or other EEG abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
EEG index value during three concentrations of nitrous oxide | During induction of anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Kate Leslie, MD, Principal Investigator — Melbourne Health
Locations (2):
- Australia (2):
  - Swinburne University, Hawthorn, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria